CLINICAL TRIAL: NCT04990882
Title: FAPI PET/CT Imaging for Cancer: A Prospective Interobserver Agreement Study
Brief Title: FAPI PET/CT Prospective Interobserver Agreement
Acronym: AGREE-FAPI
Status: Completed | Type: Observational
Sponsor: University Hospital, Essen (Other)
Responsible Party: Principal Investigator, PD Dr. med. Wolfgang Fendler, Principal Investigator, University Hospital, Essen
Other Study IDs: AGREE-FAPI
Record Dates: First submitted 2021-07-16; First posted 2021-08-05 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Malignant Neoplasm
Keywords: FAPI; cancer; Positron-Emission-Tomography; FAP; fibroblast; imaging; PET; Interobserver agreement
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Low Experience Group: Nuclear medicine physicians or radiologists with a prior experience with 68Ga-FAPI PET/CT of less than 30 studies.
  Interventions: Other: Interpretation of FAPI-PET/CT scans
- Intermediate Experience Group: Nuclear medicine physicians or radiologists with a prior experience with 68Ga-FAPI PET/CT of more than 30 studies and less than 300 studies.
  Interventions: Other: Interpretation of FAPI-PET/CT scans
- High Experience Group: Nuclear medicine physicians or radiologists with a prior experience with 68Ga-FAPI PET/CT of more than 300 studies.
  Interventions: Other: Interpretation of FAPI-PET/CT scans

INTERVENTIONS:
Other: Interpretation of FAPI-PET/CT scans — Each observer's Group will be asked to review FAPI-PET/CT scans of patients with representative cancer types.

SUMMARY:
The aim of the present study is to evaluate the interobserver agreement for FAPI PET/CT interpretations of representative cancer types and compare findings among readers with different levels of experience.

DETAILED DESCRIPTION:
Fibroblast activation protein (FAP) is expressed by many cancer-associated fibroblasts, having a pivotal role in many desmoplastic tumor histotypes (sarcoma, pancreatic cancer, colorectal cancer). 68Ga-FAPI inhibitor (FAPI) is a promising novel molecular imaging tracer for positron emission tomography with computed tomography (PET/CT), with favorable initial results in different tumor entities. Compared to 18F-FDG, 68Ga-FAPI PET/CT shows a similar biodistribution, with less background tracer uptake in the brain, oral mucosa and liver, thus making this tracer potentially suitable to detect tumor lesions in these regions.

Moreover, the FAPI ligand contains a DOTA peptide which makes it appropriate also for therapeutic options if linked with 177Lutetium or 90Yttrium.

There is an increasing number of trials aimed to assess the efficacy and the clinical impact of 68Ga-FAPI PET/CT. Therefore, the inter-observer agreement and variability with 68Ga-FAPI PET/CT need to be established.

ELIGIBILITY:
Inclusion criteria:

Nuclear medicine physicians or radiologists with a prior experience with 68Ga-FAPI PET/CT from high-volume centers (Essen, Germany; Bologna, Italy; Los Angeles, USA; Munich, Germany, Münster, Germany ) will be prospectively recruited as research observers. Each observer will be asked to report the number of previous clinical 68Ga-FAPI PET/CT scans and then will be classified on the basis of the experience in these three groups:

* Low experience (< 30 prior 68Ga-FAPI PET/CT studies);
* Intermediate experience (30 to 300 studies);
* High experience (> 300 studies) At least three observers will be needed for each group.

Exclusion criteria:

No prior PET/CT experience.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Each recruited observer will be asked to review 50 68Ga-FAPI PET/CT scans of patients with different types of tumor.
  Observers will be blinded to clinical data except of the following patient information: sex, age (years), weight (Kg), injected dose (MBq), uptake time (min), type of cancer and PET/CT indication (e.g. staging, re-staging after surgery, evaluation after therapy).
  Each observer will be also asked to record maximum standardized uptake value (SUVmax) for one exemplary lesion for each tissue (organ, node, bone).
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Agreement among observer groups in interpreting FAPI PET/CT scans | 3 Months
  Number of concordant scans among observer groups. Each scan will be rated as positive, negative or suspicion. For each scan all definite and suspicious lesions will be reported as well. Observer's reports data will be compared with an Expert Reading, which includes lesion validation, if applicable (i.e. imaging, laboratory, histopathology).

SECONDARY OUTCOMES:
Agreement among observer groups in interpreting TNM stage and semi-quantitative values. | 3 Months
  Number of concordant scans for TNM staging and for semi-quantitative values among observer groups. For each scan all definite and suspicious lesions with uptake values will be reported and a post-analysis TNM staging will be performed. Observer's reports data will be compared with an Expert Reading, which includes lesion validation, if applicable (i.e. imaging, laboratory, histopathology).

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Fendler, MD, Principal Investigator — Study Principal Investigator
Locations (1):
- Department of Nuclear Medicine, Essen, Germany

IPD SHARING:
Plan to Share IPD: No